CLINICAL TRIAL: NCT06249776
Title: Gravity Stent-Retriever System For Reperfusion Of Large Vessel Occlusion Stroke Trial (GRASSROOT)
Brief Title: Gravity Stent-Retriever System For Reperfusion Of Large Vessel Occlusion Stroke Trial
Acronym: GRASSROOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gravity Medical Technology, INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMT-GRASSROOT-24-01
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases
Keywords: Mechanical thrombectomy; Brain; Brain clot; Brain infarction; Cerebral ischemia; Neurovascular intervention; Revascularization; Reperfusion; Stent retriever; Supernova; Stroke; Gravity Medical Technology
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supernova revascularization device (Experimental): Mechanical thrombectomy with Supernova Stent Retriever
  Interventions: Device: Supernova revascularization device

INTERVENTIONS:
Device: Supernova revascularization device — Mechanical Thrombectomy

SUMMARY:
The study aims to evaluate the safety and efficacy of the Supernova stent retriever device, developed by Gravity Medical Technology, for treating acute ischemic stroke. The device is used to remove blood clots and restore blood flow to the brain .

ELIGIBILITY:
Inclusion Criteria:

1. New focal neurologic deficit consistent with being of acute cerebral ischemia origin.
2. Age 18-85 years old (inclusive).
3. Interventionalists estimate that treatment with the Supernova (first deployment in target vessel) can be achieved within 24 hours of symptom onset.
4. Intravenous thrombolysis may be given as per national guidelines and patients receiving or not receiving intravenous thrombolysis will both be eligible for inclusion in the study.
5. Admission NIH Stroke Scale score of 8-25
6. No known significant pre-stroke disability (pre-stroke mRS 0 or 1).
7. Catheter angiographic confirmation of large vessel occlusion in the intracranial internal carotid artery, the M1 or M2 segments of the middle cerebral artery, or the basilar artery that is accessible to the Supernova device.
8. For strokes in the anterior circulation, the following imaging criteria should also be met:

   1. MRI criterion: volume of diffusion restriction visually assessed ≤50 mL, OR
   2. CT criterion: ASPECTS 6 to 10 on baseline NCCT
9. Anticipated life expectancy of at least 6 months.
10. A signed informed consent by the patient or a Legally Authorized Representative or independent physician in case of oral consent.

Exclusion Criteria:

1. Subject already participating in another study of an investigational treatment device or treatment.
2. Use any other intra-arterial recanalization drug or device prior to the use of Supernova (Supernova is not the first-choice device).
3. Angiographically evident excessive arterial tortuosity precluding device access to the thrombus.
4. For all patients, severe sustained hypertension with SBP >220 and/or DBP >120; for patients treated with IV tPA, sustained hypertension despite treatment with SBP >185 and/or DBP > 110.
5. Glucose < 50 mg/dl (2.78 mmol/L) or > 400 mg/dl (22.20 mmol/L).
6. Known hemorrhagic diathesis.
7. Coagulation factor deficiency or oral anti-coagulant therapy with an international normalized ratio (INR) of more than 3.0.
8. Treatment with heparin within 48 h with a partial thromboplastin time more than two times the laboratory normal.
9. Patients who have received a direct thrombin inhibitor within the last 48 hours; must have a partial thromboplastin time (PTT) less than 1.5 times the normal to be eligible.
10. Platelet count of less than 50,000/ µL.
11. History of severe allergy to contrast medium, nickel, or Nitinol.
12. Intracranial hemorrhage.
13. Significant mass effect with midline shift.
14. Intracranial tumor (apart from small meningioma, ≤ 2 cm in diameter).
15. Stenosis or any occlusion in the deployment site or in a proximal vessel requiring treatment or preventing device access to the thrombus (for example, stenosis or occlusion in the cervical internal carotid artery or common carotid artery).
16. Presence of intracranial atherosclerotic disease requiring rescue therapy (for example, intracranial stenting).
17. Females who are pregnant or breastfeeding.
18. Known current use of narcotic drugs at the time of treatment.
19. Prior recent stroke in the past 3 months.
20. Renal failure with serum creatinine >3.0 or Glomerular Filtration Rate (GFR) <30.
21. Known cerebral vasculitis.
22. Rapidly improving neurological status defined as the improvement of greater than 8 points on the NIHSS or improvement to NIHSS of < 6 prior to the procedure.
23. Clinical symptoms are suggestive of bilateral stroke or stroke in multiple territories.
24. Ongoing seizure due to stroke.
25. Evidence of active systemic infection.
26. Known cancer with metastases.
27. Suspicion of aortic dissection, septic embolus, or bacterial endocarditis.
28. Evidence of dissection in the extra or intracranial cerebral arteries.
29. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation or anterior/posterior circulation).
30. Aneurysm in the target vessel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Successful reperfusion | Day 0 (end of procedure)
  Rate of successful reperfusion, defined as modified Thrombolysis in Cerebral Ischemia (mTICI) grade of 2b or higher
  Grade 0: No reperfusion Grade 3: Complete reperfusion
Symptomatic intracranial hemorrhage | sICH measured within 24 (18-36) hours of the study procedure
  Safety (Rate of symptomatic intracranial hemorrhage (sICH) as measured by the SITS-MOST criteria) The SITS-MOST definition of SICH is a local or remote type II parenchymal haemorrhage within 22 to 36 hours after treatment (or sooner) associated with a ≥ fourpoint deterioration on the NIHSS score from baseline or from the lowest score from baseline to 24 hours, or leading to death.
All-cause mortality | All-cause mortality measured at 90 (±14) days
  Safety (All-cause mortality)

SECONDARY OUTCOMES:
Percentage of participants with a modified Rankin Scale (mRS) score of ≤2 | 90 (±14) days post-treatment
  Effectiveness
  (The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead)
Successful Reperfusion at First Pass | Assessed at first pass of the intervention during the procedure
  Effectiveness (Successful reperfusion defined as mTICI 2b or better at first pass)
Asymptomatic Intracranial Hemorrhage | Day 1 (within 24 hours (18-36 hours) of the procedure)
  Safety (Incidence of any asymptomatic intracranial hemorrhage post-procedure)
Neurological Deterioration | Day 1 (within 24 hours (18-36 hours) of the procedure)
  Safety (defined as a ≥4-point increase in the National Institutes of Health Stroke Scale (NIHSS) score)

CONTACTS AND LOCATIONS:
Overall Officials: Dileep R. Yavagal, MD, MBBS, Study Chair — University of Miami & Jackson Memorial Hospitals
Locations (11):
- India (9):
  - Marengo CIMS Hospital, Ahmedabad, Gujarat
  - P.D. Hinduja Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Dr Balabhai Nanavati Hospital, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry
  - Yashoda Hospitals, Secunderabad, Hyderabad, Telangana
  - Yashoda Hospitals, Somajiguda, Hyderabad, Telangana
  - Apollo Hospitals, Hyderabad, Telangana
  - The Calcutta Medical Research Institute, Kolkata, West Bengal
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yavagal DR, Gaikwad SB, Vibha D, Narayan SK, Nagarajan K, Kesavarupu SR, Sharma MK, Sharaf R, Vankayalapati S, Mehta A, Das D, Doshi D, Oak P, Salunkhe M, Jankowitz B, Rai AT, Brown SB, Zaidi SF, Asif KS, Liebeskind DS, Jovin TG, Pandian J, Jadhav AP, Atchaneeyasakul K, Desai S, Giragani S; GRASSROOT Trial investigators; GRASSROOT trial investigators GRASSROOT Trial investigators. Mechanical thrombectomy for acute ischemic stroke in a low- and middle-income country: primary outcomes from the GRASSROOT Trial. J Neurointerv Surg. 2025 Dec 10:jnis-2025-024470. doi: 10.1136/jnis-2025-024470. Online ahead of print. PMID 41371775